CLINICAL TRIAL: NCT05350839
Title: Reliability and Validity of HHIRS General Quality of Life Questionnaire in Urdu Speaking Population of Pakistan
Brief Title: Reliability and Validity of HHIRS General Quality of Life Questionnaire
Acronym: HHIRS-GQOL
Status: Completed | Type: Observational
Sponsor: Helping Hand Institute of Rehabilitation Sciences (Other)
Responsible Party: Principal Investigator, Keramat Ullah, Principal HHIRST/ Chairman HHREC, Helping Hand Institute of Rehabilitation Sciences
Other Study IDs: Rec.Letter/St./2021/20/03/01
Record Dates: First submitted 2021-04-15; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Musculoskeletal Pain; Neurological Disorder
Keywords: Reliability; Validity; HHIRS-General-QOL; questionnaire; patient reported outcome measure
MeSH Terms: conditions — Musculoskeletal Pain; Nervous System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Quality of life is conceded by copious musculoskeletal and neurogenic conditions which are evaluated by manifold questionnaires. These questionnaires are obtainable in English and many other languages but in Pakistan, these cannot be applied due to differences in languages, lifestyles, culture, and activities of daily living (ADL's). In relation to the culture of Pakistan, there are many accomplishments such as offer prayers and other domestic obligation which cannot be executed appropriately if any Musculoskeletal and neurogenic disorders are existing. All these disorders can be assessed appropriately by questionnaires previously accessible but not in a single tool.

DETAILED DESCRIPTION:
HHIRS developed a general quality of life questionnaire in the Urdu language for the expediency of patients. Relation of the questionnaire with upper limb has been identified but there is no clear relation with other body regions. Consequently, the purpose of this research is to evaluate the validity and reliability of the HHIRS-General-QOL Questionnaire in the Urdu Speaking Population of Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* participants able to read and write Urdu
* neurological disorders
* musculoskeletal pain
* systemic diseases

Exclusion Criteria:

* communication disorder
* cognitive disorder

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: study population targeted will be the Urdu-speaking population with any neurological or musculoskeletal pain/ disorder impacting their quality of life.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
validity of HHIRS general quality of life questionnaire | 2 months
  validity of questionnaire will be determined by comparing the responses of patients for HHIRS-GQOL questionnaire with GHQ-12 questionnaire
Reliability of HHIRS general quality of life questionnaire | 72 hours
  reliability will be measured by comparing the score the score of questionnaires collected at two different occasions

CONTACTS AND LOCATIONS:
Overall Officials: keramat Ullah Keramat, Principal Investigator — HHIRS Trust
Locations (1):
- Helping hand Institute of Rehabilitation Sciences Trust, Mansehra, KPK, Pakistan